CLINICAL TRIAL: NCT00382343
Title: Antibiotic Prophylaxis After Acute Pyelonephritis for Prevention of Urinary Tract Infections in Children With Vesico-Ureteral Reflux.
Brief Title: A Randomized Controlled Trial on Antibiotic Prophylaxis in Children With Vesico-Ureteral Reflux
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC 35/00
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pyelonephritis; Renal Scars
Keywords: Prevention; Pyelonephritis; Renal scars; Vesico-ureteral reflux; Dimercaptosuccinic acid renal scan (DMSA)
MeSH Terms: conditions — Pyelonephritis; Vesico-Ureteral Reflux | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sulfamethoxazole/trimethoprim (Experimental): Antibiotic prophylaxis with sulfamethoxazole/trimethoprim [1-2 mg/kg trimethoprim and 5-10 mg/kg sulfamethoxazole once daily]; in case of intolerance (leucopoenia) and for children younger than 6 months: nitrofurantoin [2 mg/kg once daily]
  Interventions: Drug: Sulfamethoxazole/trimethoprim
- No prophylaxis (No Intervention)

INTERVENTIONS:
Drug: Sulfamethoxazole/trimethoprim — Sulfamethoxazole/trimethoprim prophylaxis
  Arms: sulfamethoxazole/trimethoprim

SUMMARY:
The aim of this study is to assess the effectiveness of antibiotic prophylaxis in preventing pyelonephritis and in avoiding the appearance of new scars in a sample of children under 36 months with vesico-ureteral reflux (VUR).

DETAILED DESCRIPTION:
In recent years, the effectiveness of continuous antibiotic prophylaxis in children with vesico-ureteral reflux (VUR) has been intensely discussed. The question is not only whether antibiotics are effective in preventing recurrent urinary tract infections (UTI), but also whether they alter the natural history of disease and help to prevent the appearance of new kidneys scars. The evidence on the effectiveness of antibiotic prophylaxis is scanty: randomised controlled trials (RCT) published until now are poorly designed and carried out in very heterogeneous samples of children, i.e. spanning from 6 months to 14-18 years of age and pooling patients with and without VUR. A recently updated Cochrane Systematic Review concludes that high quality RCTs are needed to determine the effectiveness of long-term antibiotics for the prevention of UTIs in susceptible children. Moreover, the presence of VUR has not been firmly shown to be a risk factor for recurrence of pyelonephritis, and a direct association between VUR and the presence of scars or the appearance of new scars has not been demonstrated; there is just an association between VUR of grade IV-V and prenatal renal dysplasia, almost exclusively in male infants. In spite of this uncertainty, several practice guidelines recommend long term antibiotic prophylaxis in children with different degrees of VUR.

The aim of this study is to assess the effectiveness of antibiotic prophylaxis in preventing pyelonephritis and in avoiding the appearance of new scars in a sample of children under 36 months with VUR.

Comparison: In a multicentre trial, 100 patients with VUR diagnosed with cystourethrography after a first episode of acute pyelonephritis or for prenatal evidence of pyelectasia will be assigned randomly to receive prophylaxis or not. Randomization will be carried out using a centralized minimization procedure to balance for sex, age group and VUR grade.

ELIGIBILITY:
Inclusion Criteria:

* presence of vesico-ureteral reflux (VUR) grade II, III or IV, based on the International Classification, mono or bilateral, diagnosed between one day and 30 months of age after a first episode of acute pyelonephritis, or after birth during diagnostic procedures planned as a consequence of prenatal ultrasonographic evidence of pyelectasia.

Exclusion Criteria:

* previous episodes of urinary tract infection (UTI), even if only suspected (e.g. an episode of fever treated with antibiotics without performing urine culture);
* VUR grade I, because of the high probability of rapid spontaneous resolution;
* VUR grade V, as requested by the Technical Scientific Committee, concerned by the high incidence of associated renal dysplasia;
* recurrence of acute pyelonephritis before the first dimercaptosuccinic acid (DMSA) renal scan, if this was positive for scars.

Ages: 1 Day to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 1999-11; Primary Completion 2003-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Recurrence of pyelonephritis | up to 4 years after enrollment
  Urinalysis and urine culture performed at each episode of fever or when symptoms of UTI occurred (eg, change in the smell of urine, anorexia, irritability)

SECONDARY OUTCOMES:
Renal scars | 4 years after enrollment
  DMSA renal scan
Persistence of vesico-ureteral reflux | 4 years after enrollment
  Cystourethrography and renal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pennesi, MD, Principal Investigator — Institute of Child Health IRCCS Burlo Garofolo, Trieste, Italy
Locations (7):
- Italy (7):
  - Sant'Orsola Hospital, Bologna, Bologna
  - Bufalini Hospital, Cesena, Cesena
  - San Polo Hospital, Monfalcone, Gorizia
  - Santa Maria degli Angeli Hospital, Pordenone, Pordenone
  - Institute of Child Health IRCCS Burlo Garofolo, Trieste, Trieste
  - San Daniele Hospital, San Daniele, Udine
  - Sant'Antonio Abate Hospital, Tolmezzo, Udine

REFERENCES:
- [Result] Pennesi M, Travan L, Peratoner L, Bordugo A, Cattaneo A, Ronfani L, Minisini S, Ventura A; North East Italy Prophylaxis in VUR study group. Is antibiotic prophylaxis in children with vesicoureteral reflux effective in preventing pyelonephritis and renal scars? A randomized, controlled trial. Pediatrics. 2008 Jun;121(6):e1489-94. doi: 10.1542/peds.2007-2652. Epub 2008 May 19. PMID 18490378